CLINICAL TRIAL: NCT03172858
Title: A Randomized Trial of Intracervical Balloon Placement Versus Intravenous Oxytocin in Women With Prelabor Rupture of Membranes and Unripe Cervices
Brief Title: Randomized Control Trial of Intracervical Balloon Placement vs Oxytocin in Women With Term PROM and Unripe Cervices
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The IRB identified too many safety issues and the study did not move ahead.
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00203535
Record Dates: First submitted 2017-04-19; First posted 2017-06-01 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Premature Rupture of Membrane; Unfavorable Cervix
Keywords: cervical ripening; term premature rupture of membrane; intracervical balloon catheter
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intracervical Balloon Catheter Group (Experimental): The intracervical balloon catheter will be passed through the cervix either with a speculum exam or by a digital exam. Then the catheter balloon will be filled with 80 cc of sterile fluid. The catheter will be pulled to tension and taped to the patient's leg.
  Patients will have the option to IV pain medication at the time of intracervical balloon placement. The intracervical balloon will remain in place for 6 hours unless it falls out spontaneously. At the 6 hour mark, a vaginal exam will assess if the intracervical balloon has pulled through the cervix or if it needs further tension. The intracervical balloon will remain in place a maximum of 12 hours. After a maximum of 12 hours in place the intracervical balloon will be removed and oxytocin will be started per protocol.
  Interventions: Device: Intracervical balloon catheter; Drug: Oxytocin
- Immediate low-dose oxytocin infusion group (Active Comparator): At our institution the policy for oxytocin infusion is to start at a low dose of 2mu/min and to increase by 2mu/min at 15 to 20 minute intervals based on how often uterine contractions are occuring. A specific order from a physician is required to increase the oxytocin dose above 20 mu/min. Oxytocin will be titrated per usual protocol.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Device: Intracervical balloon catheter — cervical ripening balloon
  Arms: Intracervical Balloon Catheter Group
Drug: Oxytocin — medication used to induce contractions

SUMMARY:
This study is designed to determine if an intracervical balloon catheter (IBC) is better than oxytocin for induction of labor in the setting of premature rupture of membranes (PROM) or breaking the bag of water prior to onset of labor. The investigators suspect that an intracervical balloon catheter will shorten the time interval from initiation of induction of labor to delivery.

DETAILED DESCRIPTION:
There are not enough studies to support the use of intracervical balloon catheter (IBC) in term prelabor rupture of membranes (PROM). Prospective randomized studies comparing IBC placement to oxytocin use in induction of labor for term PROM do not exist. Intracervical Balloon Catheter has been shown to reduce duration of labor for women with intact membranes undergoing induction of labor. The practice at this institution is to use oxytocin to start contractions when a woman has PROM. This study will examine IBC compared to oxytocin use in term PROM. This will allow for the evaluation of a cervical ripening method for term PROM that may improve women's outcomes. Other outcomes for this study are rates of infection during labor, cesarean section, and adverse maternal and/or neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

Nulliparous women, Women aged 18-50 years, Singleton gestation, Vertex presentation, Live fetus, Rupture of membranes confirmed by sterile speculum examination > 37 weeks of gestation at time of rupture of membranes, Bishop score < 6

Exclusion Criteria:

Multiparous women, Bishop score >6, Multifetal gestation, Contraindication to labor including placenta previa , Maternal fever prior to randomization: T >100.4 F , Known fetal anomalies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Time from start of induction defined as time of IBC (intracervical balloon catheter) placement or initiation of oxytocin until delivery in hours | 24-48 hours/duration of induction of labor
  length of induction

SECONDARY OUTCOMES:
Length of first stage of labor | delivery (from initial cervical dilation to 10 cm cervical dilation])
  length of first stage of labor
Cesarean delivery rate | 24-48 hours/duration of induction of labor
  number of cesarean deliveries
chorioamnionitis | 24-48 hours/duration of induction of labor
  Maternal temperature >100.4 F during labor with associated maternal or fetal tachycardia
Endometritis | from time of delivery until 2 days after delivery for vaginal deliveries and 3 days after delivery for cesarean sections
  temperature >100.4 F in the postpartum period with initiation of antibiotics in postpartum period
Postpartum hemorrhage | at time of delivery and up to 24 hours after delivery
  Estimated blood loss (EBL) >500 cc from a vaginal delivery and EBL >1000 cc from a cesarean delivery
Epidural use | 24-48 hours/duration of induction of labor
  epidural anesthesia use during labor
Neonatal 5-minute Apgar score | 5 minutes after delivery
  apgar score at 5 minutes of life after delivery of neonate
Neonatal umbilical arterial and venous acid base status | at the time of delivery
  assessment of acid-base status of neonate at the time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Whitney You, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hannah ME, Ohlsson A, Farine D, Hewson SA, Hodnett ED, Myhr TL, Wang EE, Weston JA, Willan AR. Induction of labor compared with expectant management for prelabor rupture of the membranes at term. TERMPROM Study Group. N Engl J Med. 1996 Apr 18;334(16):1005-10. doi: 10.1056/NEJM199604183341601. PMID 8598837
- [Background] Bond DM, Middleton P, Levett KM, van der Ham DP, Crowther CA, Buchanan SL, Morris J. Planned early birth versus expectant management for women with preterm prelabour rupture of membranes prior to 37 weeks' gestation for improving pregnancy outcome. Cochrane Database Syst Rev. 2017 Mar 3;3(3):CD004735. doi: 10.1002/14651858.CD004735.pub4. PMID 28257562
- [Background] Mackeen AD, Walker L, Ruhstaller K, Schuster M, Sciscione A. Foley catheter vs prostaglandin as ripening agent in pregnant women with premature rupture of membranes. J Am Osteopath Assoc. 2014 Sep;114(9):686-92. doi: 10.7556/jaoa.2014.137. PMID 25170038
- [Background] Cabrera IB, Quinones JN, Durie D, Rust J, Smulian JC, Scorza WE. Use of intracervical balloons and chorioamnionitis in term premature rupture of membranes. J Matern Fetal Neonatal Med. 2016 Mar;29(6):967-71. doi: 10.3109/14767058.2015.1027191. Epub 2015 Sep 25. PMID 25845274
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264